CLINICAL TRIAL: NCT02536807
Title: Minimally Invasive Volume Augmentation of Papillae Around Implant Restorations With Hyaluronic Acid Injection. A Randomized Controlled Clinical Trial With 6 Months Follow-up
Brief Title: Minimally Invasive Volume Augmentation of Papillae Around Implant Restorations With Hyaluronic Acid Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Malmö University (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Andreas Stavropoulos, Professor & Chair, Department of Periodontology, Malmö University
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 42297
Record Dates: First submitted 2015-08-27; First posted 2015-09-01 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2015-09

CONDITIONS: Interdental Papilla Augmentation
MeSH Terms: interventions — Hyaluronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hyaluronan (Experimental): Hyaluronan gel injection
  Interventions: Drug: Hyaluronan
- Control (Placebo Comparator): Control placebo gel injection
  Interventions: Drug: Hyaluronan

INTERVENTIONS:
Drug: Hyaluronan — HA gel injection
  Other Names: HA

SUMMARY:
Open gingival embrasures, also called "black triangles", may occur after surgical intervention or tooth replacement by an implant. They are perceived as anaesthetic by most patients and causing functional and phonetic problems. The aim of the present study is to assess the effect of injection of hyaluronic acid for papilla augmentation next to an implant restoration in a clinical controlled double-blinded randomized trial with 6 months follow-up.

DETAILED DESCRIPTION:
Background Open gingival embrasures, also called "black triangles", may occur after surgical intervention or tooth replacement by an implant. They are perceived as anaesthetic by most patients and causing functional and phonetic problems. Although micro-surgical approaches in oral surgery have considerably improved, reconstruction of a missing papilla to close an open gingival embrasure is still amongst the most challenging surgical scenarios. None of the so far reported surgical interventions are predictable. Recently, injection of hyaluronic acid, an important component of the extracellular matrix, was introduced as a minimally invasive, simple, non-surgical method to augment missing papilla tissue. Yet, controlled clinical studies on the effect of hyaluronic acid to reconstruct a missing papilla are not available so far.

Aim The aim of the present study is to assess the effect of injection of hyaluronic acid for papilla augmentation next to an implant restoration in a clinical controlled double-blinded randomized trial with 6 months follow-up.

Materials and methods Forty patients seeking treatment for open gingival embrasures next to an implant restoration will be included. Patients will be randomly assigned to test group (n=20; injection of hyaluronic acid, Hyadent Barrier Gel, BioScience, Germany; CE certificated for Europe) or control group (n=20; injection of saline solution as a placebo control medium). The following clinical parameters will be assessed at baseline and after 1, 3, and 6 months: Modified papilla index score, distance between papilla tip and contact point, area and volume of black triangle, tissue texture and colour, probing depth, clinical attachment level, presence of plaque and/or bleeding on probing, aesthetic satisfaction of the patient and the examiner and sensation during injection. At baseline and after 6 months the distance between contact point and most cervical region of the alveolar bone crest will be assessed on periapical radiographs.

ELIGIBILITY:
Inclusion Criteria:

* atrophic papillae in the maxilla or mandible anteriorly to 1st premolar next to an implant
* at least 18 years of age and adequate plaque control (full mouth plaque score < 20%)

Exclusion Criteria:

* open contact point, positive bleeding on probing and/or probing depth >5mm,
* presence of a labial recession (depth >3mm) at the neighboring teeth
* <2mm keratinized tissue at the gingival margin of the neighboring teeth/implant
* known systemic healing disorders (e.g. uncontrolled diabetes, malignancy, disease affecting connective tissue metabolism)
* regular intake of medications with an effect on mucosal healing (e.g. steroids)
* pregnancy or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
distance between papilla tip and contact point | 6 months

SECONDARY OUTCOMES:
Probing pocket depth | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- School of Dentistry, Malmö University, Malmo, Sweden